CLINICAL TRIAL: NCT06961305
Title: Post-Marketing, Prospective, Multicentre, Single-Arm, Open-Label Investigation of Alexa Medium for Correction of Lip Volume Loss Within Accepted Cosmetological Practice
Brief Title: A Post-Marketing Study of Alexa Medium for Сorrection of the Lips Volume Loss
Acronym: ALMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute Hyalual GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL-MED/REG-21
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Lip Volume Enhancement; Lip Augmentation; Aesthetic
Keywords: Aesthetic; Lip Volume; Alexa Medium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm: Alexa Medium (Experimental): Participants received one or two injections of Alexa Medium, a cross-linked hyaluronic acid gel, into the mucous membrane of the lips for aesthetic correction of lip volume loss. The second injection was optional and performed at the discretion of the investigator during the second visit.
  Interventions: Device: Cross-linked Hyaluronic Acid Gel

INTERVENTIONS:
Device: Cross-linked Hyaluronic Acid Gel — This intervention involves the injection of Alexa Medium, a sterile, cross-linked hyaluronic acid gel (17.5 mg/mL). The gel is administered into the mucous membrane of the lips for aesthetic restoration of lip volume loss. The product is supplied in a pre-filled 1 mL syringe and injected by a trained medical professional. One or two injections were administered per participant, with the second injection performed at the investigator's discretion at Visit 2. The device is manufactured by Diaco Biofarmaceutici S.r.l., Italy.

SUMMARY:
This post-marketing, prospective, multicentre, single-arm, open-label clinical investigation aimed to evaluate the safety, tolerability, and effectiveness of the injectable medical device Alexa Medium (based on cross-linked hyaluronic acid) for the correction of lip volume loss. Participants received one or two injections of the product, and effectiveness was assessed using the Global Aesthetic Improvement Scale (GAIS) and the Medicis Lip Fullness Scale (MLFS). Safety data were collected at each visit. The study demonstrated high effectiveness and safety, with most subjects achieving their personal aesthetic goals.

ELIGIBILITY:
Inclusion Criteria:

* Subject's age 25 to 70.
* Subject will receive an injection of the medical device 'Alexa Medium' manufactured by Diaco Biofarmaceutici S.r.l., Italy for correction of the lips volume loss within accepted cosmetological practice.
* Subject's lips requiring correction of the lips volume loss according to the Investigator's judgement.
* The subject has established a realistic aesthetic improvement goal that the Investigator agrees is achievable, i.e., have realistic expectations of aesthetic results.
* Subject willing to have photographs of the face taken.
* Subject psychologically able to understand the Investigation related information and to give a written informed consent.
* Subject able and agreeing to follow Investigation procedures, instructions and likely to complete all required visits.
* The subject agreed to participate in the Investigation and signed the Informed Consent Form.

Exclusion Criteria:

* Subject's age less than 25 or more than 70.
* Subject tends to develop hypertrophic scarring.
* Subjects has known hypersensitivity to cross-linked hyaluronic acid.
* Subjects has history of severe and/or multiple allergies.
* Subjects has history of herpetic rash.
* Subject has impaired haemostatic function.
* Subject is on anticoagulant medication(s) or is using substances that can prolong bleeding.
* Subject has present or past history of autoimmune disease or autoimmune deficiency.
* Subject is undergoing immunosuppressive therapy.
* Subject has acute rheumatic fever with heart complications.
* Subject has tumour in area of the IMD application.
* Subject has active tuberculosis.
* Subject with presence of any other chronic disease that in the opinion of the Investigator may interfere with the outcome of the Investigation.
* Subject is a pregnant or breastfeeding women.
* Subject is presenting with cutaneous inflammatory and/or infectious diseases (acne, herpes, etc.) in area of the IMD application.
* Subject plans laser correction, deep chemical peels or dermabrasion during the potential participation in this Investigation.
* Subject has undergone recently laser correction, deep chemical peels, dermabrasion or surface peels, so the inflammatory reaction from the peel is significant.
* Subject has a permanent implant in the area of the IMD application.
* Subject has already injected more than 18 mL of dermal fillers per 60 kg of body mass per year.
* Subject refuses or is suspected of inability to comply with the requirements of the CIP.
* Subject has difficulty understanding the language in which the informed consent is written.
* Any other reason that the Investigator believes prevents the subject from participating in the Investigation (including suspicion of body dysmorphic disorder).
* Subject takes part in the other Investigation.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Global Aesthetic Improvement Scale (GAIS) Score at Day 60 | Day 60 ±5 days
  Change in GAIS score from baseline to Day 60, as evaluated by the Investigator. GAIS is a 5-point scale ranging from 1 (exceptional improvement) to 5 (worsened patient).
Medicis Lip Fullness Scale (MLFS) Score at Day 60 | Day 60 ±5 days
  hange in MLFS score from baseline to Day 60, as evaluated by the Investigator. MLFS is a 5-grade scale (1=very thin lips, 5=very full lips)

CONTACTS AND LOCATIONS:
Locations (4):
- Poland (3):
  - Provita Sp. z o.o., Katowice
  - Ośrodek medyczny OSTEOMED s.c., Krakow
  - Ostrowieckie Centrum Medyczne, Ostrowiec Świętokrzyski
- Institute Hyalual LLC, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided